CLINICAL TRIAL: NCT05132920
Title: Fight INflammation to Improve Outcome After Aneurysmal Subarachnoid HEmorRhage
Acronym: FINISHER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Pharmacy of the University Hospital Leipzig- AöR (Unknown); nextevidence GmbH (Unknown)
Responsible Party: Principal Investigator, Erdem Güresir, MD, Prof. Dr. Erdem Güresir, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCH-201803; 2021-000732-54 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): 3 x 8 mg (2 ml) dexamethasone daily for days 1-7 and 1 x 8 mg (2 ml) dexamethasone daily for days 8-21 in addition to aneurysm treatment and best medical intensive care of SAH patients
  Interventions: Drug: Dexamethasone
- Control arm (Placebo Comparator): 3 x 2 ml Placebo daily for days 1-7 and 1 x 2 ml Placebo daily for days 8-21 in addition to aneurysm treatment and best medical intensive care of SAH patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 3 x 8 mg dexamethasone daily for days 1-7 and 1 x 8 mg dexamethasone daily for days 8-21
  Arms: Experimental arm
Drug: Placebo — 3 x 2 ml Placebo daily for days 1-7 and 1 x 2 ml Placebo daily for days 8-21
  Arms: Control arm

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a fatal disease with high morbidity and mortality. While the primary injury results from the initial bleeding and cannot be influenced, secondary injury through vasospasms and delayed cerebral ischemia (DCI) during the course of the disease might be a target for intervention in order to improve outcome. To date, beside the aneurysm treatment to prevent re-bleeding and the administration of oral nimodipine, there is no causal therapy available, so that novel treatment concepts are desperately needed. There are strong indications that inflammation contributes to DCI and therefore poor outcome and plays a major role in SAH. Some studies suggest a beneficial effect of anti-inflammatory drugs like glucocorticoids (GC) in SAH patient, but there are no data from randomized controlled trials proving or disproving the beneficial effect of GC, so that current guidelines do not recommend the use of GC in SAH so far.

This multi-center trial aims to generate the first confirmatory data in a controlled randomized fashion that dexamethasone (DEX) improves the outcome in a clinically relevant endpoint in SAH patients. Moreover, this trial will generate first data in a secondary analysis, whether the initial inflammatory state of SAH patients defines a subgroup that particularly responds to a treatment with DEX.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, equal or older than 18 years old
2. Written consent to participate in the study by the patient or his legal representative (emergency inclusion by next of kin or consultant physician under the responsibility of the principal investigator is possible)
3. Confirmed diagnosis of aneurysmal SAH and onset within 48 hours before inclusion.

Exclusion Criteria:

1. SAH due to any other cause than aneurysm rupture (e.g. traumatic, arteriovenous malformation (AVM), fistula, dissection)
2. Any condition that, in the judgement of the Investigator, could impose hazards to the patient if study therapy is initiated or affects the participation of the patient in the study
3. Patients with obvious evidence of irreparable brainstem or thalamic injury
4. Patients with foreseeable difficulties to attend follow-ups adequately
5. Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in this clinical trial
6. Current positive pregnancy test (e.g. β-HCG test in serum)
7. Known history of hypersensitivity to the investigational drug or to drugs with a similar chemical structure
8. Severe infectious diseases
9. Known angle-closure or open angle glaucoma
10. Known ulceration in the gastro-intestinal tract
11. History of gastro-intestinal bleeding
12. Long-term treatment with corticosteroids prior SAH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) at 6 months after SAH | 6 months
  Dichotomized modified Rankin Scale (mRS) 6 months after subarachnoid haemorrhage. The dichotomization will be done in the classes "favourable" (mRS 0-3) versus "unfavourable " (mRS 4-6) outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Güresir, Prof. Dr., Principal Investigator — Department of Neurosurgery, University Hospital Leipzig
Locations (13):
- Germany (13):
  - Eberhard Karls University of Tübingen, Tübingen, Baden-Wurttemberg
  - University of Ulm/BKH Günzburg, Günzburg, Bavaria
  - Klinikum rechts der Isar, School of Medicine, Technical University of Munich, München, Bavaria
  - University Medical Center Regensburg, Regensburg, Bavaria
  - Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main, Hesse
  - Hannover Medical School, Hanover, Lower Saxony
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University of Cologne, Cologne, North Rhine-Westphalia
  - University Hospital of Essen, Essen, North Rhine-Westphalia
  - University Hospital Leipzig, Leipzig, Saxony
  - Otto von Guericke University Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité-Universitätsmedizin Berlin, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Derived] Guresir E, Lampmann T, Bele S, Czabanka M, Czorlich P, Gempt J, Goldbrunner R, Hurth H, Hermann E, Jabbarli R, Krauthausen M, Konig R, Lindner D, Malinova V, Meixensberger J, Mielke D, Nemeth R, Darkwah Oppong M, Pala A, Prinz V, Rashidi A, Roder C, Sandalcioglu IE, Sauvigny T, Schebesch KM, Timmer M, Vajkoczy P, Wessels L, Wild F, Wilhelm C, Wostrack M, Vatter H, Coch C. Fight INflammation to Improve outcome after aneurysmal Subarachnoid HEmorRhage (FINISHER) trial: Study protocol for a randomized controlled trial. Int J Stroke. 2023 Feb;18(2):242-247. doi: 10.1177/17474930221093501. Epub 2022 May 3. PMID 35361026